CLINICAL TRIAL: NCT04253392
Title: Research to Further Inform Thinking About the Role of LINX for Reflux Disease
Brief Title: RETHINK REFLUX Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: TRX_2018_01
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux Disease; GERD; Reflux; Regurgitation; Esophageal Disease; Lower Esophageal Sphincter; LES; Magnetic Sphincter Augmentation; MSA
MeSH Terms: conditions — Gastroesophageal Reflux; Esophageal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: LINX Reflux Management System — The LINX Reflux Management System consists of a series of titanium beads each with a magnetic core connected with independent titanium wires to form an annular shape when implanted. The attractive force of the magnetic beads is designed to provide additional strength to keep a weak lower esophageal sphincter (LES) closed. During swallowing, the magnetic beads slide away from each other on the independent titanium wire "links" to allow esophageal distention as the bolus passes by.
  Other Names: LINX

SUMMARY:
The RETHINK REFLUX Registry is a post-market prospective, multi-center, observation, single arm, long-term safety surveillance registry of subjects implanted with the LINX device. The primary objective of the study is to confirm the long-term safety profile of the LINX device and procedure (implant/explant) up to 10 years post-implant.

DETAILED DESCRIPTION:
The RETHINK REFLUX Registry or Research to further inform thinking about the role of LINX for Reflux Disease is sponsored by Ethicon Endo-Surgery, Inc. This is a post-market prospective, multi-center, observational, single arm, long-term safety surveillance registry of subjects implanted with the LINX device. Up to 500 subjects will be enrolled and implanted at up to 50 centers in both the US and selected countries outside the US with regulatory approval for the LINX Reflux Management System. The study will collect data from patients 10 years post implant. The primary objective of the study is to confirm the long-term safety profile of the LINX device and procedure (implant/explant). Secondary objectives include Effectiveness, Health Economics and Health Utilization.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is >or=21 years old
2. Subject with prospective plans for a LINX procedure
3. Subject provides written informed consent
4. Subject must be willing and able to complete questionnaires/ surveys electronically (ePROs)

Exclusion Criteria:

1. Subject who was previously implanted with LINX device
2. Any reason which the Principal Investigator believes may cause the subject to be non-compliant with or unable to meet the protocol requirements (i.e. medical illness and/or limited life expectancy of less than 10 years)

Note: Physicians should refer to the LINX Reflux Management System IFU for a complete list of contraindications, warnings, and precautions.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients successfully implanted (treated) with the LINX Reflux Management System for the treatment of GERD (Implant success defined as leaving the surgical suite with a device in situ)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2032-07-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse Events | 10 years
  Adverse events related to the LINX device and/or procedure (implant/explant) limited to:
  * All related serious adverse events
  * All related adverse events of dysphagia and or odynophagia requiring treatment (only)
  * LINX migration
  * LINX erosion
Safety - Explant/Removal | 10 years
  LINX explant/removal
Safety - Hiatal Hernia Reoccurrence | 10 years
  Hiatal hernia requiring repair (occurring after the LINX implant)

SECONDARY OUTCOMES:
Effectiveness | 10 years
  Follow-up questionnaires Gastroesophageal Reflux Disease Esophageal Health Related Quality of Life Questionnaire (GERD-HRQL), Foregut Symptoms Questionnaire (FSQ) and GERD Medication Survey] will be collected and compared to baseline with evaluation to include:
  1. Percentage of subjects reporting >or=50% reduction in GERD-HRQL scores
  2. Percentage of subjects reporting the following on the FSQ:
     * Elimination of moderate or severe regurgitation
     * Reduction in extra-esophageal symptoms
     * Maintain the ability to belch
     * Maintain the ability to vomit
  3. Percentage of subjects reporting > or = 50% reduction in average daily proton pump inhibitor (PPI) use
Health Economics - Work Productivity and Activity Impairment | 10 years
  Measure of the impact of GERD on a subject's ability to work will be collected through the responses on the Work Productivity and Activity Impairment (WPAI) questionnaire. Percentages of impairment at baseline will be compared to scores collected annually. Four types of scores will be analyzed:
  * Absenteeism (work time missed)
  * Presenteeism (impairment of work/ reduced on-the-job effectiveness)
  * Work productivity loss (overall work impairment/ absenteeism plus presenteeism)
  * Activity impairment
Health Economics - GERD Treatment Decision-Making Process (Subject's Perspective) | Baseline
  To better understand a subject's process for making GERD related healthcare decisions and his/her care pathways, the LINX Interest Survey will be collected once at baseline, prior the implant procedure
Health Economics - Healthcare Utilization | 10 years
  Analysis of healthcare economics in subjects who seek treatment for worsening of GERD symptoms and device/procedural complications over 10 years. A Healthcare Encounter Survey will be completed by subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Tomaszewski, MD, Study Director — Ethicon Endo-Surgery
Locations (28):
- United States (21):
  - University of South Alabama, Mobile, Alabama
  - NW Allied Bariatric and Foregut Surgery, Tucson, Arizona
  - Keck Hospital of USC, Los Angeles, California
  - Institute of Esophageal and Reflux Surgery, Englewood, Colorado
  - University of Southern Florida (Tampa General Hospital), Tampa, Florida
  - OSF Medical Group, Peoria, Illinois
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Sparrow Hospital / Sparrow Medical Group, Lansing, Michigan
  - East Carolina University / Vidant Medical Center, Greenville, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Gen Surg Assoc / Fairfield Medical Center, Lancaster, Ohio
  - Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Minimal Access Surgery/Prisma Health - Upstate, Greenville, South Carolina
  - Adv Surg Assoc / Self Regional Healthcare, Greenwood, South Carolina
  - Lexington Surgery, West Columbia, South Carolina
  - Panhandle Weight Loss Center, Amarillo, Texas
  - Houston Methodist, Houston, Texas
  - Bariatric Medical Institute of Texas, San Antonio, Texas
  - Richmond Surg / Henrico Doctors' Hospital, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Fox Valley Surgical Associates, Appleton, Wisconsin
- MedUni Wien / Universitatsklinik fur Chirurgie, Vienna, Austria
- Marien Hospital Herne, Herne, Germany
- Univ of Milano / IRCCS Policlinico San Donato, San Donato Milanese, Italy
- National University Hospital, Singapore, Singapore
- United Kingdom (3):
  - Epsom Hospital, Epsom
  - Guy's and St. Thomas' Hospitals, London
  - RefluxUK, Royal Tunbridge Wells

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu.